CLINICAL TRIAL: NCT00312338
Title: Topical Treatment of Bacterial Conjunctivitis and Its Effect on Microbial Flora
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Collaborators: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single
Other Study IDs: CMS-05-11
Record Dates: First submitted 2006-04-04; First posted 2006-04-10 (Estimated); Results first posted 2010-02-02 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2010-02

CONDITIONS: Bacterial Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Bacterial | interventions — Moxifloxacin

ARMS (2):
- Infected Patient treated with Vigamox (Experimental): Conjunctivitis-Infected Patient receiving Vigamox 0.5% in both eyes three times daily for 7 days.
  Interventions: Drug: VIGAMOX
- Healthy Subjects (No Intervention): Healthy Subjects receiving no treatment

INTERVENTIONS:
Drug: VIGAMOX — 1 drop of VIGAMOX® ophthalmic solution 0.5% in both eyes TID for 7 days
  Arms: Infected Patient treated with Vigamox

SUMMARY:
Topical Treatment of Bacterial Conjunctivitis and its Effect on Microbial Flora

ELIGIBILITY:
Inclusion Criteria:

* Patients from 1 to 13 years of age that have diagnosis of bacterial conjunctivitis in either or both eyes (for < 3 days duration) based on clinical observation; matched healthy controls

Exclusion Criteria:

* Cannot have had bacterial conjunctivitis symptoms as reported by parent for > 2 days

Ages: 1 Year to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 137 (Actual)
Dates: Start 2006-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J. Lichtenstein, M.D., Principal Investigator — Investigator / Contact
Locations (1):
- Multiple Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment started in June 2006 and ran until January 29 2008. The study sites included three sites (AZ, CA and IL)
Pre-assignment Details: No specific pre-assignment activities.
Groups:
- Infected Patients: Infected Patients
- Healthy Subjects: Healthy Subjects
Period: Overall Study
Arm/Group | Infected Patients | Healthy Subjects
Started | 105 | 57
Completed | 83 | 54
Not Completed | 22 | 3
Not completed — Adverse Event | 7 | 2
Not completed — Lost to Follow-up | 9 | 1
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Subsequent infection | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infected Patients | Healthy Subjects | Total
Number analyzed (Participants) | 105 | 57 | 162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 105 | 57 | 162
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 28 | 76
  Male | 57 | 29 | 86

OUTCOME MEASURES:

1. Primary Outcome: Susceptability Changes in Streptococcus Pneumoniae Distal to the Site of Instillation
Description: Susceptibility change refers to a change in vulnerability of a specified bacterial strain to antibiotic treatment. Susceptibility was assessed by broth microdilution methods recommended by the Clinical and Laboratory Standards Institute (CLSI).
  0% = zero isolates were resistant to antibiotic 100% = all isolates were resistant to antibiotic
Time Frame: Day 0 and Day 42
Measure: Number; unit: Percent of resistant isolates
Arm/Group | Infected Patients | Healthy Subjects
Number analyzed (Participants) | 83 | 54
Percent of resistant isolates
  Day 0 | 0 | 0
  Day 42 | 0 | 0

2. Primary Outcome: Susceptability Changes in Staphylococcus Aureus Distal to the Site of Instillation
Description: as for outcome 1
Time Frame: Day 0, Day 42
Measure: Number; unit: Percent of resistant isolates
Arm/Group | Infected Patients | Healthy Subjects
Number analyzed (Participants) | 83 | 54
Percent of resistant isolates
  Day 0 | 8.3 | 0
  Day 42 | 0 | 0

3. Primary Outcome: Susceptability Changes in Haemophilus Influenzae Distal to the Site of Instillation
Description: as for outcome 1
Time Frame: Day 0, Day 42
Measure: Number; unit: Percent of resistant isolates
Arm/Group | Infected Patients | Healthy Subjects
Number analyzed (Participants) | 83 | 54
Percent of resistant isolates
  Day 0 | 0 | 0
  Day 42 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 0 to Day 42
Arm/Group | Infected Patients | Healthy Subjects
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/57
Other Adverse Events (participants affected / at risk) | 6/105 | 0/57
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infected Patients (N=105) | Healthy Subjects (N=57)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 0 (0)

LIMITATIONS AND CAVEATS:
Limited source documents.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less